CLINICAL TRIAL: NCT06995976
Title: Dosimetry and Preliminary Clinical Application Study of a Novel Probe Targeting CD73
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-CD73
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Malignant Tumour
MeSH Terms: conditions — Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-dPNE PET/CT (Experimental): Intravenous injection of 68Ga-dPNE. 68Ga-dPNE PET/CT will be used to detect tumors.
  Interventions: Drug: 68Ga-dPNE
- 18F-FDG PET/CT (Experimental): Intravenous injection of 18F-FDG. 18F-FDG PET/CT will be used to detect tumors.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 68Ga-dPNE — Intravenous injection of 68Ga-dPNE. 68Ga-dPNE PET/CT will be used to detect tumors.
  Arms: 68Ga-dPNE PET/CT
Drug: 18F-FDG — Intravenous injection of 18F-FDG.18F-FDG PET/CT will be used to detect tumors.
  Arms: 18F-FDG PET/CT

SUMMARY:
As a new CD73-targeted PET radiotracer, 68Ga-dPNE, is promising as an excellent imaging agent applicable to various cancers. In this study, we observed the safety, biodistribution and radiation dosimetry of 68Ga-dPNE in human volunteers. Furthermover, we conducted a comparative analysis of 68Ga-dPNE and 18F-FDG imaging to assess both the radiation dosimetry and diagnostic efficacy of 68Ga-dPNE.

DETAILED DESCRIPTION:
The boom in radiopharmaceuticals continues to persist, including their driving effects in the field of immunotherapy. CD73 (ecto-5'-nucleotidase), a key purine metabolic enzyme, catalyzes the conversion of extracellular nucleotides to adenosine, promoting tumor immune evasion and unfavorable clinical outcomes. Notably, CD73 is highly expressed in 74.3% of breast cancer cases, with its prevalence exceeding 45% in liver, gastric, colorectal, and ovarian cancers. As a new CD73-targeted PET radiotracer, 68Ga-dPNE, is promising as an excellent imaging agent applicable to various cancers. The present study aimed to evaluate the biodistribution, pharmacokinetics, and dosimetry of 68Ga-dPNE, and performed a head-to-head comparison with 18F-FDG PET/CT scans in patients with various cancers.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent and be able to follow up.

Exclusion Criteria:

Pregnant or lactational women; who suffered from severe hepatic and renal insufficiency.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
SUV of tumors | Through study completion, an average of 3 months
  Compare the SUV of tumors between 68Ga-dPNE PET/CT and 18F-FDG PET/CT.

SECONDARY OUTCOMES:
Diagnostic value | Through study completion, an average of 3 months
  Sensitivity and specificity of 68Ga-dPNE in patients with various types of cancer and compare it with 18F-FDG PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No